CLINICAL TRIAL: NCT07257575
Title: A Phase II Randomized Controlled Clinical Study of Serplulimab Combined With Chemotherapy in the Treatment of Patients With Locally Advanced Gastric Adenocarcinoma
Brief Title: A Randomized Controlled Study of Serplulimab Combined With Chemotherapy for Locally Advanced Gastric Adenocarcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPACE-neo
Record Dates: First submitted 2025-03-10; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer Stage III
Keywords: local advanced gastric cancer; neoadjuvant chemotherapy; PD-1 inhibitor; FLOT
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel)+Serplulimab (Experimental)
  Interventions: Drug: FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel)+Serplulimab
- FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel) (Active Comparator)
  Interventions: Drug: FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel)

INTERVENTIONS:
Drug: FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel)+Serplulimab — The subjects will first receive four cycles of neoadjuvant FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel) combined with serplulimab treatment, administered once every two weeks (Q2W). Imaging assessments will be conducted after the completion of the 2nd and 4th cycles of neoadjuvant therapy, followed by standard surgery. Postoperatively, they will continue with four cycles of adjuvant chemotherapy based on fluoropyrimidine combined with serplulimab, starting 4-6 weeks after surgery.
  Arms: FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel)+Serplulimab
Drug: FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel) — The subjects will first receive four cycles of neoadjuvant FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel) treatment, administered once every two weeks (Q2W). Imaging assessments will be conducted after the completion of the 2nd and 4th cycles of neoadjuvant therapy, followed by standard surgery. Postoperatively, they will continue with four cycles of adjuvant chemotherapy based on fluoropyrimidine, starting 4-6 weeks after surgery.
  Arms: FLOT (Fluorouracil+Leucovorin+Oxaliplatin+Docetaxel)

SUMMARY:
The goal of this clinical trial is to learn if FLOT chemotherapy combined with serplulimab can improve the pathological complete response (pCR) rate in patients with stage III gastric cancer. The main question it aims to answer is:

Can FLOT chemotherapy combined with serplulimab improve the pathological complete response (pCR) rate in patients with stage III gastric cancer? Researchers will compare serplulimab with a blank control group to see if it can improve the pathological complete response (pCR) rate in patients with stage III gastric cancer.

Participants will :

Receive serplulimab combined with FLOT chemotherapy or FLOT chemotherapy alone every 2 weeks Undergo imaging assessments at 4 weeks and 8 weeks Undergo surgery based on imaging results after 8 weeks Receive postoperative serplulimab combined with adjuvant chemotherapy or adjuvant chemotherapy alone

DETAILED DESCRIPTION:
Gastric cancer (GC) remains a major global health challenge, with approximately 1 million new cases and 650,000 deaths reported annually in recent years. The incidence rate of GC is significantly higher in Asia, particularly in South Korea and China. Specifically, according to the 2020 statistics from the International Agency for Research on Cancer (IARC), China accounts for 44% of global incident cases and 48.6% of global mortality cases related to gastric cancer, respectively. Furthermore, in 2022, China recorded 358,700 new gastric cancer cases and 260,400 deaths annually. The overall survival rate and median survival time of Chinese GC patients were 33.53% and 28.68 months, respectively.

In recent years, perioperative treatment has remained a research hotspot in the field of gastric cancer. Prior to the advent of the immunotherapy era, a two-drug combination regimen (SOX regimen: oxaliplatin plus S-1) served as the primary standard of care across East Asia. Notably, findings from the RESOLVE study have established the SOX regimen as one of the standard treatment options for the perioperative management of gastric cancer in China. In contrast, based on the outcomes of the FLOT4-AIO study, the FLOT regimen has long been the cornerstone of perioperative chemotherapy for gastric cancer in Western countries. More recently, the MATTERHORN study integrated immunotherapy into the perioperative treatment landscape, with results demonstrating that the addition of immunotherapy to the FLOT regimen further significantly improves event-free survival (EFS) and overall survival (OS). The success of this pivotal study has revolutionized our understanding of perioperative immunotherapy, and the FLOT-immunotherapy combination has now gained widespread acceptance in clinical practice.

Serplulimab is a monoclonal antibody with demonstrated safety and favorable clinical efficacy across multiple cancer types. Therefore, the objective of this clinical trial is to evaluate whether FLOT chemotherapy combined with serplulimab can enhance the pathological complete response (pCR) rate in patients with stage III gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Have a full understanding of the study and voluntarily sign the Informed Consent Form (ICF);
2. The tumor is located in the stomach, pathologically confirmed as adenocarcinoma, with clinical stage III (cT3-4aN1-3M0) determined by enhanced CT/MRI examination;
3. Tumor specimens show PD-L1 positivity (CPS ≥ 1). At the time of enrollment, there must be sufficient tumor tissue available for assessing PD-L1 expression levels (subjects undergoing repeated screening do not need additional PD-L1 testing);
4. No restriction on gender, aged 18-70 years;
5. Generally in good condition, with an ECOG performance status of 0-1, and no contraindications to surgery;
6. Physical condition and organ function allow for major abdominal surgery;
7. Expected survival ≥ 3 months;
8. Laboratory test results within 7 days prior to enrollment must meet the following criteria:

   1. WBC > 3.50 × 10⁹/L and < 9.50 × 10⁹/L, ANC > 1.5 × 10⁹/L, Hb ≥ 80 g/L, PLT ≥ 100 × 10⁹/L;
   2. Serum bilirubin ≤ 1.5 × ULN, AST and ALT ≤ 2.5 × ULN;
   3. Creatinine ≤ 1.5 × ULN or serum clearance > 60 ml/min;
   4. INR and aPTT ≤ 1.5 × ULN (for subjects not receiving anticoagulation therapy); subjects receiving anticoagulants must be on a stable dose;
9. Demonstrates good compliance and is able to cooperate with the study protocol's laboratory, auxiliary examinations, and relevant specimen collection;
10. Women of childbearing potential (including those in menopause due to chemotherapy or other medical reasons) must agree to use contraception from the time of signing the ICF to at least 5 months after the last dose of study treatment or concurrent chemotherapy (whichever is later). They must also agree not to breastfeed during this period. Men must agree to use contraception from the initiation of the study drug to at least 7 months after the last dose of study drug or concurrent chemotherapy (whichever is later).

Exclusion Criteria:

1. HER2-positive status, defined as IHC3+ or IHC2+ with FISH+; or known MSI-H/dMMR.
2. Tumor involvement of the esophagogastric junction (EGJ).
3. Known allergy to citric acid monohydrate, sodium citrate dihydrate, mannitol, or polysorbate (components of the investigational drug).
4. History or concurrent diagnosis of other malignancies (excluding completely resected basal cell carcinoma, stage I squamous cell carcinoma, carcinoma in situ, mucosal carcinoma, superficial bladder cancer, or any other cancer with no recurrence for at least 5 years).
5. Uncontrolled pericardial effusion, pleural effusion, ascites, gastrointestinal bleeding, or high bleeding risk within 2 weeks prior to enrollment.
6. Weight loss exceeding 20% within 2 weeks prior to enrollment.
7. Inability to take oral medication.
8. History of chemotherapy, radiotherapy, immunotherapy, or surgery for gastric cancer.
9. Previous treatment with anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies (or any other antibody targeting T-cell co-stimulatory or checkpoint pathways).
10. Tyrosine kinase inhibitor treatment within 2 weeks prior to enrollment.
11. Long-term use of immunosuppressive drugs or systemic/local corticosteroids at immunosuppressive doses (e.g., >10 mg/day prednisone or equivalent).
12. Vaccination with any anti-infective vaccine (e.g., influenza, varicella) within 4 weeks prior to enrollment.
13. Uncontrolled systemic diseases, such as diabetes or hypertension.
14. Current or required anticoagulant therapy (except for low-dose aspirin used as antiplatelet therapy).
15. Active autoimmune diseases or history of autoimmune diseases (e.g., interstitial pneumonitis, uveitis, colitis, hepatitis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; exceptions include vitiligo or childhood asthma resolved without intervention; patients requiring bronchodilators for asthma are excluded).
16. Active tuberculosis (TB), ongoing anti-TB treatment, or anti-TB treatment within 1 year prior to screening.
17. History of lung diseases confirmed by imaging (preferably CT) or clinical results, such as interstitial pneumonia, non-infectious pneumonia, pulmonary fibrosis, or acute lung diseases.
18. Contraindications to oxaliplatin, docetaxel, 5-FU, or leucovorin.
19. Pregnant or breastfeeding women, or women who might be pregnant.
20. Active hepatitis.
21. Positive test results for any of the following: HIV-1 antibody, HIV-2 antibody, HTLV-1 antibody, or HCV antibody.
22. Any clinically significant disease or condition deemed by the investigator to affect protocol compliance, the ability to sign the informed consent form (ICF), or suitability for participation in this clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
pCR rate | Perioperative
  pathological complete regression rate

SECONDARY OUTCOMES:
MPR rate | Perioperative
R0 resection rate | Perioperative
OS | 5 years
EFS | 5 years
perioperative complication rate | Up to postoperative 30 days
Chemotherapy-related side effects | At the end of each cycle of chemotherapy (each cycle is 14 days)

CONTACTS AND LOCATIONS:
Locations (1):
- No. 106, Zhongshan 2nd Road, Yuexiu District, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No